CLINICAL TRIAL: NCT00989209
Title: Improvement of Facial Symmetry With Myofunctional Therapy Combined to Botulinum Toxin Injections in Long Standing Facial Paralysis
Brief Title: Myofunctional Therapy in Facial Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Paula Nunes Toledo, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAPPesq 890/04
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2009-10-05 (Estimated); Status verified 2009-10

CONDITIONS: Facial Paralysis
Keywords: facial paralysis; asymmetry; myofunctional therapy; botulinum toxin; facial evaluation
MeSH Terms: conditions — Facial Paralysis | interventions — Botulinum Toxins, Type A; Myofunctional Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: myofunctional prior to botulinum (Active Comparator): All the facial paralysis patients received treatment with botulinum toxin type A to the non-paralyzed side, according to the Institution Protocol. To the participants of Group A, botulinum toxin was applied after myofunctional therapy.
  Interventions: Drug: Botulinum Toxin Type A; Procedure: myofunctional therapy
- B: myofunctional after botulinum (Active Comparator): All the facial paralysis patients received treatment with botulinum toxin type A to the non-paralyzed side, according to the Institution Protocol. To the participants of Group B, botulinum toxin was applied before myofunctional therapy.
  Interventions: Drug: Botulinum Toxin Type A; Procedure: myofunctional therapy

INTERVENTIONS:
Drug: Botulinum Toxin Type A — All the patients received a one-time treatment with botulinum toxin type A to the non-paralyzed side, according to the Institution Protocol,the total dose used per patient ranged from 15-69U, mean 37.9±5.4U.
  Other Names: BOTOX (Allergan)
Procedure: myofunctional therapy — All the patients were submitted to individual myofunctional therapy with the speech therapist, once a week, by four weeks.The myofunctional therapy began with isometric maneuvers for muscular elongation on the non paralyzed side, and on the paralyzed side when microsurgical reconstruction was present. It also included isotonic maneuvers to increase muscle tonus and isokinetic maneuvers to increase force on the paralyzed side.

SUMMARY:
Objective: Quantify the benefits of myofunctional therapy associated to botulinum toxin injection in patients with long standing facial unilateral palsy.

DETAILED DESCRIPTION:
Twenty-five patients with long standing facial palsy were studied; all had been previously treated for facial reanimation. Patients were randomly divided in two groups; Group A did the myofunctional therapy sessions with the speech therapist before the botulinum toxin injection, while the participants of Group B did the myofunctional therapy after it.

ELIGIBILITY:
Inclusion Criteria:

* facial paralysis with more than 2 years elapsed since the onset of symptoms
* surgically treated for reanimation at least 12 months before
* static and/or dynamic facial asymmetry causing aesthetic concern

Exclusion Criteria:

* spastic paralysis
* serious systemic or neuromuscular diseases
* cognition impairment
* pregnant women

Ages: 16 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2005-01; Primary Completion 2005-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Clinical score | 2 months

SECONDARY OUTCOMES:
Facial Disability Index (self-report instrument) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra G Salles, Study Director — University of Sao Paulo General Hospital; Marcus C Ferreira, Study Chair — University of Sao Paulo General Hospital; Paula N Toledo, Principal Investigator — University of Sao Paulo General Hospital; Claudia F Andrade, Study Director — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Salles AG, Toledo PN, Ferreira MC. Botulinum toxin injection in long-standing facial paralysis patients: improvement of facial symmetry observed up to 6 months. Aesthetic Plast Surg. 2009 Jul;33(4):582-90. doi: 10.1007/s00266-009-9337-9. Epub 2009 Mar 28. PMID 19330369